CLINICAL TRIAL: NCT04297085
Title: Prospective Cohort Study on the Determinants of Venous THromboembolic Recurrence. BREIZH-Cohorte
Brief Title: Prospective Cohort Study on the Determinants of Venous THromboembolic Recurrence
Acronym: BREIZH-Cohorte
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BREIZH-Cohorte (29BRC19.0304)
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-12

CONDITIONS: Thromboembolic Venous Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cases (Experimental)
  Interventions: Biological: Biologic sample

INTERVENTIONS:
Biological: Biologic sample — Biological samples will be taken from the subjects included

SUMMARY:
The main objective of the BREIZH-Cohorte study is to determine the incidence of recurrent short, medium and long-term thromboembolic venous disease as well as risk factors for recurrence in two specific populations: patients under 50 years of age, men and women (5 year recurrence), as well as cancer patients (all ages) (1 year recurrence).

DETAILED DESCRIPTION:
Deep vein thrombosis (DVT) and pulmonary embolism (PE) are two clinical manifestations of the same entity, thromboembolic venous disease. This disease is frequent: the annual incidence of thromboembolic venous disease estimated between 1 and 2 cases per 1000 inhabitants per year in France, comparable to that observed in North America. This disease is potentially serious: the mortality from PE, the most severe manifestation of thromboembolic venous disease (one third of PE for two thirds of DVT) is 10% at 3 months, twice as high as that of myocardial infarction. However, the risk of PE in isolated DVT is major (more than 50% of cases). Thus, whether it is a PE or a DVT, anticoagulant treatment, a cornerstone of therapeutic management, must therefore be initiated urgently, without waiting for the results of diagnostic confirmatory examinations.

The major complications occurring after a thromboembolic venous disease are venous thromboembolic recurrence (VTE) and the long-term consequences: post-thrombotic syndrome and the development of post-embolic pulmonary hypertension. VTE recurrence has significant mortality, particularly in the form of PE (15%, compared to 2% in the form of DVT). As for long-term complications of VTE, about 20-30% of patients with DVT develop post-thrombotic syndrome at 5 years (27), while 0.15% to 5% of patients with PE develop post-embolic pulmonary hypertension at 1 year.

While major progress has been made over the past 20 years in terms of diagnosis, primary and secondary prevention, identification of risk factors for VTE and prognostic factors, however, two particular subgroups deserve to be specifically investigated: young subjects, whether women (hormonal exposure) or men (often idiopathic thromboembolic venous disease), and cancer patients. In the latter, the progress made on anti-cancer treatments is helping to modify the data on the risk of VTE as well as the duration of treatment of VTE in these patients.

Thus, this prospective cohort covers two subgroups of patients with thromboembolic venous disease: young subjects (≤50 years) or those who have cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 or over, or a minor with the consent of the parents and the minor, presenting with a thromboembolic venous disease
* 50 and under or any age if active cancer
* Affiliated to social security
* Accepting to participate in the study.

Exclusion Criteria:

* Inability to communicate (comprehension disorder).
* Refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2020-05-28 (Actual); Primary Completion 2050-04 (Estimated); Study Completion 2050-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of thromboembolic venous disease | 20 years
  Recurrence of thromboembolic venous disease will be established at the end of patient monitoring

SECONDARY OUTCOMES:
Haemorrhages under anticoagulant | 20 years
  Haemorrhages under anticoagulant will be identified during patient follow-up
Mortality | 20 years
  Mortality will be identified during patient follow-up
Arterial complications | 20 years
  Arterial complications will be identified during patient follow-up
Long-term complications | 20 years
  long-term complications (chronic thrombo-embolic pulmonary hypertension, chronic thrombo-embolic disease) will be identified during patient follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francis COUTURAUD, MD, PHD, Principal Investigator — EA3878 (GETBO), Brest University Hospital in France
Locations (4):
- France (4):
  - CHRU Brest, Brest
  - HIA Clermont Tonnerre Brest, Brest
  - CH Morlaix, Morlaix
  - CH de Cornouaille, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.